CLINICAL TRIAL: NCT02099656
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Bronchoscopy Study to Evaluate the Effects of Lebrikizumab on Airway Eosinophilic Inflammation in Patients With Uncontrolled Asthma on Inhaled Corticosteroids and a Second Controller Medication
Brief Title: A Study Evaluating the Effects of Lebrikizumab on Airway Eosinophilic Inflammation in Participants With Uncontrolled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB29260; 2014-000275-14 (EudraCT Number)
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lebrikizumab (Experimental): Participants with uncontrolled asthma on ICS therapy (not specified in the protocol) and a second controller medication, will receive SC injection of lebrikizumab on Days 1 and 8, and on Weeks 4 and 8.
  Interventions: Drug: Lebrikizumab; Drug: Inhaled corticposteroids (ICS); Drug: Second Asthma Controller Medication
- Placebo (Placebo Comparator): Participants with uncontrolled asthma on ICS therapy (not specified in the protocol) and a second controller medication, will receive SC injection of lebrikizumab matching placebo on Days 1 and 8, and on Weeks 4 and 8.
  Interventions: Drug: Placebo; Drug: Inhaled corticposteroids (ICS); Drug: Second Asthma Controller Medication

INTERVENTIONS:
Drug: Lebrikizumab — Lebrikizumab will be administered by SC injection on Day 1, Day 8, Week 4, and Week 8.
  Other Names: RO5490255
  Arms: Lebrikizumab
Drug: Placebo — Lebrikizumab matching placebo will be administered by SC injection on Day 1, Day 8, Week 4, and Week 8.
  Arms: Placebo
Drug: Inhaled corticposteroids (ICS) — Participants will continue their ICS controller therapy, as they are receiving prior to screening, throughout the study. Protocol does not specify any particular ICS.
Drug: Second Asthma Controller Medication — Participants will continue their asthma controller therapy, as they are receiving prior to screening, throughout the study.

SUMMARY:
This Phase II, randomized, double-blind, placebo-controlled, multicenter study will evaluate the effects of lebrikizumab on airway eosinophilic inflammation in participants with uncontrolled asthma who are using inhaled corticosteroid (ICS) treatment and a second controller medication. Enrolled participants will undergo a 3-week screening period during which assessments, including a bronchoscopy procedure, will be made. Participants will subsequently be randomized to receive lebrikizumab or placebo by subcutaneous (SC) injection on Day 1, Day 8, Week 4, and Week 8. Participants will continue their standard of care therapy throughout the study. End of treatment assessments will be taken at Week 12. Total study period, including screening and follow-up, is expected to last 23 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis for greater than or equal to (>/=) 12 months prior to Visit 1
* Bronchodilator response demonstrated within the 12 months before Visit 1 or at Visit 1, 2, or 3 of screening
* Pre-bronchodilator FEV1 of 40 percent (%) - 80% predicted at both Visits 2 and 3
* On ICS therapy at a total daily dose of 500-2000 mcg of fluticasone propionate dry powder inhaler (DPI) or equivalent for >/= 6 months prior to Visit 1, with no changes within 4 weeks prior to Visit 1, and no anticipated changes throughout the study
* On an eligible second controller medication (long-acting Beta-agonist [LABA), leukotriene receptor antagonist [LTRA], long-acting muscarinic antagonists [LAMAs] or theophylline) for 6 months prior to Visit 1, with no changes within 4 weeks prior to Visit 1, and no anticipated changes throughout the study
* Uncontrolled asthma at Visit 1 and/or 2 and at Visit 3
* Chest X-ray or computed tomography (CT) scan within 12 months prior to Visit 1 or chest X-ray during the screening period (prior to Visit 3) that confirms the absence of other clinically significant lung disease
* Demonstrated adherence with controller medication during the screening period

Exclusion Criteria:

* Maintenance oral corticosteroid therapy, defined as daily alternate-day oral corticosteroid maintenance therapy within 3 months prior to Visit 1
* Treatment with systemic corticosteroids within 4 weeks prior to Visit 1 or during the screening period for any reason, including an acute exacerbation event
* Any infection requiring hospital, intravenous (IV) or intramuscular (IM) antibiotic treatment or any respiratory infection within 4 weeks prior to Visit 1 or during screening. Any infection requiring oral antibiotic treatment with 2 weeks prior to Visit 1 or during screening, or any parasitic infection within 6 months prior to Visit 1 or during screening
* Active tuberculosis requiring treatment within 12 months prior to Visit 1
* Known immunodeficiency, including, but not limited to, human immunodeficiency virus (HIV) infection
* History of interstitial lung disease, chronic obstructive pulmonary disease (COPD), or other clinically significant lung disease other than asthma
* Known current malignancy or current evaluation for a potential malignancy
* Unable to safely undergo elective flexible fiberoptic bronchoscopy
* Clinically significant medical disease that is uncontrolled despite treatment, that is likely, in the opinion of the investigator, to impact the participant's ability to participate in the study, or to impact the study assessments
* History of alcohol or drug abuse that would impair or risk the participant's full participation in the study, in the opinion of the investigator
* Current smoker or history of smoking (greater than [>] 10 pack-years), or unwillingness to abstain from smoking for the duration of the study
* Past and/or current use of any anti-interleukin (IL)-13 or anti-IL-4/IL-13 therapy, including lebrikizumab
* Use of a licensed or investigational monoclonal antibody other than anti-IL-13, or anti IL-4/IL-13, including, but not limited to, omalizumab, anti-IL-5, or anti-IL-17, within 6 months or 5 drug half-lives prior to Visit 1 (whichever is longer) or during screening
* Use of a systemic immunomodulatory or immunosuppressive therapy within 3 months or 5 drug half-lives prior to Visit 1 (whichever is longer) or during screening
* Use of other investigational therapy within 4 weeks or 5 drug half-lives prior to Visit 1 (whichever is longer) or during screening
* Initiation of or increase in allergen immunotherapy within 3 months prior to Visit 1 or during screening
* Body mass index >38 kilograms per square meter (kg/m^2)
* Body weight <40 kilograms (kg)
* History of bronchial thermoplasty

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2016-10-13 (Actual)

PRIMARY OUTCOMES:
Relative Change From Baseline in the Number of Airway Submucosal Eosinophils per Surface Area of Basal Lamina (Cells per Square Millimeter [Cells/mm^2]) | From Baseline to Week 12

SECONDARY OUTCOMES:
Absolute Change From Baseline in Number of Airway Submucosal Eosinophils per Surface Area of Basal Lamina (Cells/mm^2) | From Baseline to Week 12
Relative Change From Baseline in the Number of Airway Epithelial Eosinophils per Surface Area of Basal Lamina (Cells/mm^2) | From Baseline to Week 12
Absolute Change From Baseline in Number of Airway Epithelial Eosinophils per Surface Area of Basal Lamina (Cells/mm^2) | From Baseline to Week 12
Relative Change From Baseline in Number of Airway Submucosal Eosinophils per Volume of Submucosa (Cells per Cubic Millimeter [Cells/mm^3]) | From Baseline to Week 12
Absolute Change From Baseline in Number of Airway Submucosal Eosinophils per Volume of Submucosa (Cells/mm^3) | From Baseline to Week 12
Relative Change From Baseline in Number of Airway Epithelial Eosinophils per Volume of Epithelium (Cells/mm^3) | From Baseline to Week 12
Absolute Change From Baseline in Number of Airway Epithelial Eosinophils per Volume of Epithelium (Cells/mm^3) | Form Baseline to Week 12
Change From Baseline in Blood Eosinophil Count | From Baseline to Week 12
Change From Baseline in Immunoglobulin E (IgE) Levels | From Baseline to Week 12
Change From Baseline in Serum Periostin Levels | From Baseline to Week 12
Change From Baseline in Chemokine Ligand (CCL)-13 Levels | From Baseline to Week 12
Change From Baseline in CCL-17 Levels | From Baseline to Week 12
Change From Baseline in Lung Epithelial Cell Chloride Channel Accessory 1 (CLCA1) Gene Expression | From Baseline to Week 12
Change From Baseline in Lung Epithelial Cell SerpinB2 Gene Expression at Week 12 | From Baseline to Week 12
Change From Baseline in Lung Epithelial Cell CCL-26 Gene Expression | From Baseline to Week 12
Change From Baseline in Lung Epithelial Cell Nitric Oxide Synthase 2 (NOS2) Gene Expression | From Baseline to Week 12
Change From Baseline in Lung Epithelial Cell Periostin (POSTN) Gene Expression | From Baseline to Week 12
Relative Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) | From Baseline to Week 12
Relative Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) | From Baseline to Week 12
Percentage of Participants With Treatment-Emergent Adverse Events | From Baseline to Week 20
Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Lebrikizumab | Baseline up to Week 20 (assessed at Baseline, Weeks 8 and 20/dosing termination or early termination)
Serum Lebrikizumab Concentration at Week 12 | Predose (Hour 0) at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- United States (16):
  - University of Arizona, Tucson, Arizona
  - LAC-USC Medical Center, Los Angeles, California
  - University of California Davis Health System; Division of Pulmonary and Critical Care Medicine, Sacramento, California
  - Yale School of Medicine, New Haven, Connecticut
  - University of Miami School of Medicine - Sylvester at Deerfield, Deerfield Beach, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals & Clinics; Internal Medicine, Iowa City, Iowa
  - Brigham and Women's Hospital; Pulmonary Division, Boston, Massachusetts
  - Washington University; Pediatrics, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center; Gastroenterology & Digestive Health, Winston-Salem, North Carolina
  - Pen Memory Center, Philadelphia, Pennsylvania
  - Temple University Hospital ; Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - UTMB Pathology Clinical Services, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital-SCC/WCM, Edmonton, Alberta
  - VGH Research Pavilion, Vancouver, British Columbia
  - McMaster University Health Sciences Center, Hamilton, Ontario
- France (2):
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Groupe Hospitalier Sud - Hôpital Haut Lévêque, Pessac
- Connolly Hospital, Dublin, Ireland
- Skånes Universitetssjukhus, Lund, Lund, Sweden
- United Kingdom (4):
  - Queen's University Belfast; NICRN Respiratory Research Office, Belfast
  - Glenfield Hospital, Leicester
  - St Mary's Hospital, London
  - The Medicines Evaluation Unit, Manchester

REFERENCES:
- [Derived] Austin CD, Gonzalez Edick M, Ferrando RE, Solon M, Baca M, Mesh K, Bradding P, Gauvreau GM, Sumino K, FitzGerald JM, Israel E, Bjermer L, Bourdin A, Arron JR, Choy DF, Olsson JK, Abreu F, Howard M, Wong K, Cai F, Peng K, Putnam WS, Holweg CTJ, Matthews JG, Kraft M, Woodruff PG; CLAVIER Investigators. A randomized, placebo-controlled trial evaluating effects of lebrikizumab on airway eosinophilic inflammation and remodelling in uncontrolled asthma (CLAVIER). Clin Exp Allergy. 2020 Dec;50(12):1342-1351. doi: 10.1111/cea.13731. Epub 2020 Oct 4. PMID 32909660